CLINICAL TRIAL: NCT04387253
Title: Study of Late Fetal Loss in Poitou-Charentes. GYNE-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: GYNE-COVID
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Identification of the Mother or Fetus Contamination by SARS Cov-2; Research the Presence of Viruses at Different Sites of the Mother and the Fetus or Father; The Survey Builds on a Network Work Already Organized Around the CPDPN of Poitou-Charentes; Analysis Laboratories of the Poitiers CHU

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Identification by PCR of the SARS-COV-2 virus in samples taken from the fetus — Identification by PCR of the SARS-COV-2 virus in samples taken from the fetus Presence of SARS-COV-2 virus in samples taken from mother and father. Circulating anti-SARS-COV-2 antibodies in the mother.

SUMMARY:
Maternal-fetal transmission in the second or third trimester of pregnancy of the SARS-COV-2 virus could explain some late fetal losses.

Finding a cause in the context of fetal loss is essential for parents and caregivers. It helps to understand the history of the disease, to address the possible risk of a recurrence and to plan for future pregnancies.

If the maternal-fetal transmission of COVID 19 is confirmed and that it is responsible for obstetric complications, a preventive action could be proposed to the patients by the preconception vaccination.

The investigators are seeking to clarify the frequency of this transmission is information awaited by caregivers, women, couples in particular when the latter are in distress from late fetal loss.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with late spontaneous abortion (≥15 weeks of gestation)
* Benefiting from a Social Security scheme
* Patient who consented to participate in the study
* Free subject, without tutorship, curatorship or subordination

Exclusion Criteria:

* Persons not benefiting from a Social Security scheme or not benefiting from it through a third party.
* Concurrent participation in another clinical research study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Estimate the prevalence of SARS-CoV-2 infection in women with late fetal loss of unexplained cause. | 2 months
  Identification by PCR of the SARS-COV-2 virus in samples taken from the fetus

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France